CLINICAL TRIAL: NCT03761524
Title: Evaluation of the Effect of Customized V Plate Fixation Versus a Conventional Superior -Inferior Miniplates Fixation of Mandibular Angle Fracture on Mouth Opening and Radiographical Parameters Randomized Clinical Trial
Brief Title: Evaluation of Customized V Plate Versus Conventional Miniplates of Mandibular Angle Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hiba Obad Saleh Saeed, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 543
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Mandibular Fractures
Keywords: Angle fracture; superior-inferior plate fixation; custom made plate fixation; postoperative complications
MeSH Terms: conditions — Mandibular Fractures; Postoperative Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Because the two interventions used in this trial are easily recognized by the participants and the investigator, neither the investigator nor the participant can be blinded. But, assessor and the statistician will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Customized V plate fixation (Experimental): Computed tomography (CT) scan of the Facial bones (Axial cuts, DICOM file, Gantry tilt zero and minimal thickness of 1mm )is taken for the patients and a customized V pattern plate
  Interventions: Procedure: Customized V plate fixation
- Conventional miniplates fixation (Active Comparator): Conventional superior-inferior miniplates fixation of mandibular angle fixation
  Interventions: Procedure: Conventional miniplates fixation

INTERVENTIONS:
Procedure: Customized V plate fixation — (CT) scan is taken for the patients and a customized V pattern plate will be designed .Intraoral approach will be done to expose the angle fracture.Fracture site will be exposed and reduced in normal anatomic position guided by the CAD/CAM plate. MMF will be done.Fracture fragments will be fixed using CAD/CAM plate .
  Arms: Customized V plate fixation
Procedure: Conventional miniplates fixation — Intraoral approach will be done to expose the angle fracture.Fracture site will be exposed and reduced in normal anatomic position. MMF will be done.Fracture fragments will be fixed using conventional miniplates fixation of angle fracture.
  Arms: Conventional miniplates fixation

SUMMARY:
The aim of the study to evaluate the effect of customized V pattern plate fixation versus a conventional superior-inferior mini plates fixation of mandibular angle fracture on mouth opening and radio graphical parameters.

DETAILED DESCRIPTION:
The mandibular angle is one of the most common sites for fractures, accounting for 23-42% of all cases of mandibular fractures. Moreover, mandibular angle fractures have the highest postoperative complications among all mandibular fractures, and the loosening of screws and fracturing of plates are main reasons for the complications.The most widely used treatment modality for mandibular angle fracture is the use of one miniplate fixation ,The other one uses two mini-plates, with a upper mini-plate fixed at the same place of previous treatment which corresponds to the tension band of the mandible, and the lower mini-plate fixed at the inferior border of the mandible which corresponds to the compression band of the mandible, however, based on recent experimental and clinical studies, the stability provided by the miniplate fixation of mandibular angle fractures has become a point of contention among surgeons .In order to decrease the need for plate removal, reduce the operative time and improve the stability of the fixation system, a customized V pattern plate design is an appropriate plate structure for fractured mandible using the minimum output values for stress of plate and displacement of bony segments to seek maximum reduction volume on an original plate .Patient satisfaction include: clinical parameters such are occlusion, pain, facial swelling, maximal mouth opening, sensory function, and surgical wound ,these should be evaluated postoperatively ,radio graphical evaluation is also an important parameter to assess adequate reduction of the fractured segments .

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least a unilateral unfavorable angle fracture indicated for Open reduction internal fixation alone or in combination with fracture elsewhere in the mandible or midrace.
* Patients should be free from any systemic disease that may affect normal healing of bone, and predictable outcome

Exclusion Criteria:

* Patients with systemic disease (may affect normal healing).
* Patients with old and/or malunited fractures (affect accuracy of reduction of the fractured segments).
* Patients whom cannot tolerate follow up intervals (affect accuracy of study results).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Mouth Opening | Every week for 1 month ,3 months and 6 months postoperative
  Mouth Opening is evaluated by measurement of maximal interincisal opening between maxilaary and mandibular central incisiors by the caliper and measuring unit is mm
Radiographical parameters | At 3 and 6 months postoperatively
  Radiographical parameters (Bone Density) is detected through CT scan to evaluate bone density in Hounsfield unit in the area of plate fixation to determine the effect of the plate stress over the fracture site Measures format will be summarized as mean

SECONDARY OUTCOMES:
Occlusion | immediate postoperative day
  Occlusion will be evaluated by intraoral examination and write in dental chart whether normal or abnormal occlusion

CONTACTS AND LOCATIONS:
Overall Officials: Hiba O Saleh, Phd.student, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry-Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saleh HO, Moussa BG, Salah Eddin KA, Noman SA, Salah AM. Assessment of CAD/CAM Customized V Pattern Plate Versus Standard Miniplates Fixation in Mandibular Angle Fracture (Randomized Clinical Trial). J Maxillofac Oral Surg. 2023 Dec;22(4):995-1005. doi: 10.1007/s12663-023-02027-x. Epub 2023 Oct 27. PMID 38105847